CLINICAL TRIAL: NCT03557411
Title: A Phase II Clinical Trial of SHR-1210 （an Anti-PD-1 Inhibitor） Simultaneously Combined With Hypofraction Radiotherapy in Patients With Previously Treated Oligometastatic NSCLC
Brief Title: A Trial of SHR-1210 (an Anti-PD-1 Inhibitor) in Combination With Hypofraction Radiotherapy in Patients With NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jinming Yu, Director of the hospital, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-RT-IIT-NSCLC-01
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: SHR-1210,radiotherapy,Oligometastases,NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab

STUDY DESIGN:
Intervention Model Description: SHR-1210 Simultaneously Combined with Hypofraction Radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1210 +Hypofraction radiotherapy (Experimental): SHR-1210 （an Anti-PD-1 Inhibitor） Simultaneously Combined with Hypofraction Radiotherapy
  Interventions: Drug: SHR-1210

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 （an Anti-PD-1 Inhibitor） Simultaneously Combined with Hypofraction Radiotherapy
  Other Names: Hypofraction Radiotherapy

SUMMARY:
This is a phase II clinical trial of SHR-1210 （an anti-PD-1 Inhibitor） simultaneously combined with hypofraction radiotherapy in patients with previously treated oligometastatic NSCLC.

It is a single center, single arm, open label trial. Subjects with oligometastatic non-small-cell lung cancer who is previously treated will be recruited. 12 subjects will be enrolled at the first part of the study which aims to evaluate the tolerability of SHR-1210 in combination with hypofraction radiotherapy. 30 subjects will be enrolled at the second part of the study which aims to evaluate the primary efficacy and safety of SHR-1210 in combination with hypofraction radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will voluntarily participate in this study and sign informed consent.
* NSCLC subject with 1 to 5 distant metastatic lesions in stage IV.
* No clear driven genes (including but not limited to EGFR, ALK).
* Previously received more than 1 chemotherapy regimen and progressed/recurred.
* At least one lesion is suitable for hypofraction radiotherapy.
* There is at least one measurable lesion.
* 18 to 75 years old
* ECOG 0-1
* The function of vital organs meets the following requirements. ANC≥1.5×10^9/L, PLT≥100×10^9/L, Hb≥9g/dL, ALB≥3g/dL, TSH ≤ULN, Bilirubin ≤ 1 times ULN; ALT and AST ≤1.5 times ULN. AKP ≤ 2.5 times ULN. CREA ≤1.5 times ULN or CCr≥60mL/min。
* The estimated survival period is more than 3 months.
* Female Subjects of childbearing potential must have a negative serum pregnancy test within 72 hours before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 3 months after the last dose of study treatment.

Exclusion Criteria:

* The subjects had any history of autoimmune disease or active autoimmune disease.
* Subjects are using immunosuppressive agents, or systemic, or absorptive, local hormone therapy to achieve immunosuppression.It is still in use within 2 weeks of the entry.
* Subjects with severe allergic reactions to other monoclonal antibodies.
* The subjects had a central nervous system metastases of clinical symptoms.
* Central squamous cell lung carcinoma.
* Imaging (CT or MRI) shows that tumors invade large blood vessels or are indistinct with blood vessels.
* Imaging (CT or MRI) showed significant pulmonary vacuity or necrotic tumors,Borderline adenocarcinoma accompanied by a cavity can be considered after discussion with investigator.
* Failing to properly control the clinical symptoms or disease of the heart.
* Subjects had active infections.
* Subjects may receive other systemic antitumor therapy during the study period.
* Other clinical trials of drugs were used in the first four weeks of the first medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-07-09 (Estimated); Study Completion 2020-07-09 (Estimated)

PRIMARY OUTCOMES:
Clinically significant toxicity | First cycle (28 days)
  above grade 3 AEs
6-month-PFS | From the start of treatment to 6 months.
  6-month-progression free survival rate

SECONDARY OUTCOMES:
AEs+SAEs | from the first drug administration to within 30 days for the last SHR-1210 dose
  Adverse Events and Serious Adverse Events
PFS | up to 2 years
  Progression-Free-Survival
ORR | At baseline,at the time point of every 8 weeks
  Objective Response Rate
DCR | at the time point of every 8 weeks
  Disease Control Rate
OS | up to 2 years
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: JINGMIN YU, PhD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided